CLINICAL TRIAL: NCT07166861
Title: Supporting Practices In Respecting Elders Phase 2
Brief Title: Annual Wellness Visits vs GRACE-augmented Annual Wellness Visits For Older Adults With High Needs - Phase 2
Acronym: SPIRE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brandeis University (Other); Indiana University School of Medicine (Other); Dartmouth-Hitchcock Medical Center (Other); Atrium Health Wake Forest Baptist (Other); Griffin Hospital (Other); Patient-Centered Outcomes Research Institute (Other); Baylor Scott and White Health (Other)
Responsible Party: Principal Investigator, Christine S. Ritchie, MD, MPH, Director, Center for Aging and Serious Illness, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025P000230; PLACER-2022C3-30604 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2025-07-21; First posted 2025-09-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aging; Preventive Care; Multimorbidity; Palliative Care
Keywords: annual wellness visit; geriatric collaborative care; complex care needs; geriatric assessment; implementation; comparative effectiveness
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial with 2 parallel arms. The investigators will enroll patients with complex care needs in each arm. Other participants studied will include caregivers and clinical team members.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor team will be blinded to the intervention assignments of participants. Due to the nature of the intervention, the participants, the investigator, and the care providers are unable to be blinded to the participant assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Annual Wellness Visits (AWV) (Active Comparator): Randomize 16 practices to AWV and assess impact on the population deemed by study algorithm as high-risk and recruit 90 participants from each practice (n=90/practice) to complete surveys prior to the intervention and 18 months later.
  Interventions: Other: Annual Wellness Visit
- Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE) (Experimental): Randomize 16 practices to AWV+GRACE and assess impact on the population deemed by study algorithm as high-risk and recruit 90 participants from each practice (n=90/practice) to complete surveys prior to the intervention and 18 months later.
  Interventions: Other: Annual Wellness Visit; Other: Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE)

INTERVENTIONS:
Other: Annual Wellness Visit — Completion of a structured Annual Wellness Visit (AWV) questionnaire administered by an assigned practice staff member for Medicare beneficiaries deemed by study algorithm as high-risk. Those responses will then be used by the primary care team to place any needed referrals and offer any indicated personal health advice and create a care plan for the coming year. Routine usual care from the primary care practice will occur.
  Other Names: AWV
Other: Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE) — The practice will initiate the Geriatric Resources and Assessment for the Care of Elders (GRACE) program for Medicare beneficiaries deemed by study algorithm as high-risk and meeting other study criteria (see below). After completion of the in-home structured annual wellness visit (AWV) and GRACE assessment by the NP/SW team, responses will be reviewed and applied to construct an individualized care plan using the GRACE protocols inclusive of advance care planning, health maintenance, medication management, assistance with any difficulty walking, falls, dementia, depression, chronic pain, malnutrition, weight loss, urinary incontinence, visual impairment, hearing impairment, or caregiver burden.
  Other Names: GRACE
  Arms: Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE)

SUMMARY:
This study consists of three aims focused on examining the feasibility of adding the Geriatric Resources and Assessment for the Care of Elders (GRACE) model to structured Annual Wellness Visits (AWVs) to improve patient and caregiver outcomes and reduce hospitalizations in older adults with complex health needs. The objectives are to:

1. Co-design a community-centric implementation strategy for the AWVs vs AWVs + GRACE -augmented care (AWV GRACE) study arms
2. Develop a referral pathway and algorithm to optimize enrollment of eligible participants
3. Conduct a pilot clinical trial to assess the feasibility of the AWV GRACE intervention.

DETAILED DESCRIPTION:
In the United States, 10% of patients account for half of health care costs. Many of these are older adults with complex health and social care needs (referred to as "older adults with complex needs"). They see a doctor on average 9.6 times per year, 3 times more often than older adults overall. Patients, caregivers/care partners experience care as confusing and disorganized. Clinicians in primary care practices and accountable care organization (ACO) leaders face critical dilemmas about how best to care for older adults with complex needs. Patient stakeholders providing feedback on preferred care models worry about fragmented care. Many also prefer to be at home. Evidence suggests that optimal care of older adults with complex needs involves an interprofessional team of doctors, nurses, social workers and other health care staff in partnership with patients and care partners to provide person-centered care plans, guided by evidence-based geriatric assessments. Few primary care practices provide this type of care, but Medicare ACOs and other value-based care models such as Medicare Advantage plans are well positioned to link clinicians and provide support for complex patients, their caregivers and care partners. ACOs are groups of clinicians, often housed in healthcare systems, who share in savings if they deliver high-quality care. Unlike traditional fee-for-service payment arrangements, the payment models in ACOs reward efficient, patient centered care that also minimizes unhelpful (and sometimes harmful) institutional care. ACOs are eager to optimize effective care for their patients with complex needs, but best strategies are unknown.

In 2011, to encourage value-based care, Annual Wellness Visits (AWVs) were introduced as a new Medicare Part B benefit. AWVs, as conceived by Medicare, seek to incorporate routine comprehensive assessment by primary care practices of older adults' geriatric health risks using questionnaire-based assessments completed by the patient or care partner. The goal of an AWV is to produce a Personalized Preventive Plan (PPP) for older adults. While uptake by clinicians has accelerated, uptake is lower for more vulnerable older adults. In Medicare Shared Savings Program (MSSP) Accountable Care Organizations (ACOs), an average of 55% of beneficiaries had an AWV in 2021 vs only 42% for adults 75-85 years old and dually eligible for Medicaid and Medicare.

AWVs have potential value as an organizing tool for patients and families and clinician teams as one time each year that someone looks at all aspects of care including understanding the care team, determining needed screening and preventive care, reviewing needs for assistance with activities of daily living, testing cognition, reviewing medications from multiple providers, and care coordination that can prevent acute episodes and hospitalization. For consistent and predictable impact, AWVs would be conducted systematically using evidence-based tools and structured protocols in response to patient needs elicited in AWVs. Although there is growing evidence that AWVs lead to increased screenings and reduced use of inpatient care, some are concerned that they also lead to increased use of low value testing after a visit. Furthermore, studies suggest that AWVs are underutilized in minoritized and socially vulnerable populations.

An evidence-based approach to support geriatric care planning for complex patients that offers solutions to identified problems that has been tested in primary care is the Geriatric Resources for the Assessment and Care of Elders (GRACE) program. GRACE is a protocolized inter-professional co-management model that was developed to improve the patient experience of care, provide patients and care partners with a designated point of contact in a nurse/social worker team, reduce utilization costs, and supporting overburdened primary care physicians by managing complex patients. The core components of the GRACE model include: 1) an individualized care plan developed by a nursing/social work team based on 2) an initial in-home assessment, 3) structured protocols, and 4) close co-management with the patient's primary care provider, who reviews, provides their input and endorses the plan. The care plan is built using GRACE Protocols for common geriatric conditions and providing a checklist to ensure a standardized approach to care. The care model was developed using extensive feedback from patients and family care partners. The GRACE Support Team designed it as a patient/care partner support system interfacing with the patient's primary care team to implement the care plan. In a randomized, controlled trial, patients at high risk for hospital admission who received GRACE team care versus a 'usual care' control group had decreased acute care utilization and costs with positive return on investment; improved quality of care; increased patient and provider satisfaction; and improved quality of life. However, GRACE has not been adopted by many ACOs and its additional value to the more commonly used AWV has not been established.

The purpose of the Supporting Practices in Respecting Elders (SPIRE) study is to address this gap in knowledge with the overall goal of improving the lives of older adults with complex needs cared for in primary care practices. The study will opportunistically evaluate two primary care programs aimed at improving care in older adults. The AWV is currently standard of care and is being used regularly in primary care clinics. However, AWVs is a "one size fits all" approach and may not be effective or appropriate for older adults with functional limitations and complex care needs and may not adequately meet the wellness needs of a diverse population of older adults. GRACE is an Evidence-based Practice specifically designed for older adults with complex care needs. GRACE was designed to address the health and health care challenges faced by low-income seniors with multiple chronic conditions including a comprehensive in-home assessment performed by a nurse practitioner and social worker (the GRACE Support Team). This in-home physical and social evaluation will build on the self-report AWV screening questions (promoted as the standard by CMS/Medicare) and brings together information learned at the in-home assessment back to an expanded GRACE team, which is led by a geriatrician and includes a pharmacist and mental health liaison (typically a licensed clinical social worker). No complex care delivery model such as GRACE has yet been implemented at scale. To date, health systems appear to find it easier to implement AWVs rather than AWVs augmented by GRACE in their high-need older adult populations. Therefore, a test of the comparative effectiveness of AWVs (usual care) versus AWVs augmented by GRACE will inform health system leaders and clinicians on optimal approaches for high cost, high need older adults with complex health and social needs.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 65 years or older
* Eligible for an AWV (Medicare/Medicare Advantage) during the study period
* Residential mailing address within a radius of the practice that can be achievably reached via a home visit
* English or Spanish speaking
* Be able to provide consent and / or have a proxy able to consent to study participation.
* Meet criteria for complex health care needs, by virtue of having a Probability of Repeated Admissions (PRA) score of 0.35 or greater AND/OR Kim Syndrome on Aging (efrailty indicator) score of 0.35 or greater

Caregiver Inclusion Criteria:

* Age 18 years or older
* English or Spanish speaking
* Be able to provide consent to study participation
* Be identified by an eligible patient for participation in the study

Clinician Inclusion Criteria:

* Age 18 years or older
* English or Spanish speaking
* Be able to provide consent to study participation
* Adult health professionals who work at participating ACOs and primary care practice sites (e.g. physicians, advanced practice clinicians, nurses, social workers, clinic staff.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6080 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalizations | 12, 18, and 24 months.
  Count of hospitalizations during the observation period, evaluated at the participant level.
Patient experience: Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey (CG-CAHPS) with Patient Centered Medical Home 1.0 supplement (PCMH CAHPS) | Baseline and 18 months.
  The CAHPS Clinician & Group Survey (CG-CAHPS) asks patients to report on their experiences with providers and staff in primary care and specialty care settings, using a 6 month recall period. The Patient-Centered Medical Home (PCMH) Item Set is a set of supplemental questions that is added to the adult version of the CAHPS Clinician & Group Survey (CG-CAHPS) to gather more information on patient experience with the domains of primary care that define a medical home.
  Scoring for most items is on a 4 point scale 1=never 2=sometimes 3=usually 4=Always. Minimum and Maximum scores vary with the number of items used. The Provider Rating item is on a 11 point scale from 0 to 10,where 9,10 are considered "high" scores.

SECONDARY OUTCOMES:
Physical health | Baseline and 18 months.
  PROMIS Global PH
Mental health | Baseline and 18 months.
  PROMIS Global MH
Caregiver strain | Baseline and 18 months.
  Modified Caregiver Strain Index
Clinician Well being | Baseline and 18 months.
  Professional Fulfillment Index

OTHER OUTCOMES:
Exploratory Geriatric Outcomes - Number of participants with new ICD-10 diagnosis codes | 36 months
  New ICD-10 diagnosis codes in cognitive status, physical function status or mood categories
Exploratory Geriatric Outcomes- number of participants that complete advanced care planning documents | 36 months
  Completion of health care proxy or advance care planning documents
Exploratory Geriatric Outcomes - number of participants with inappropriate medications | 36 months
  Numbers of potentially inappropriate medications

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Griffin Health, Derby, Connecticut
  - Mass General Brigham, Boston, Massachusetts
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Baylor Scott & White Health, Temple, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data can be available by request only after academic journal publication. Any formal requests should be sent by external research teams and will be reviewed by the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available upon request after academic journal publication.
Access Criteria: Access criteria will be determined and confirmed by the corresponding author upon review of the formal data request.

REFERENCES:
- [Result] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Result] Measuring hope: Development of the Herth Hope Index. Journal of Nursing Scholarship, 32, 309-315.
- [Result] Singh GK. Area deprivation and widening inequalities in US mortality, 1969-1998. Am J Public Health. 2003 Jul;93(7):1137-43. doi: 10.2105/ajph.93.7.1137. PMID 12835199
- [Result] Kind AJ, Jencks S, Brock J, Yu M, Bartels C, Ehlenbach W, Greenberg C, Smith M. Neighborhood socioeconomic disadvantage and 30-day rehospitalization: a retrospective cohort study. Ann Intern Med. 2014 Dec 2;161(11):765-74. doi: 10.7326/M13-2946. PMID 25437404
- [Result] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Result] Practice Transformation. American Medical Association. Accessed December 21, 2022. https://www.ama-assn.org/practice-management/sustainability/practice-transformation
- [Result] Maslach Burnout Inventory Manual, 4th Edition. ResearchGate. Accessed December 21, 2022. https://www.researchgate.net/project/Maslach-Burnout-Inventory-Manual-4th-Edition
- [Result] Katzan IL, Lapin B. PROMIS GH (Patient-Reported Outcomes Measurement Information System Global Health) Scale in Stroke: A Validation Study. Stroke. 2018 Jan;49(1):147-154. doi: 10.1161/STROKEAHA.117.018766. PMID 29273595
- [Result] Thornton M, Travis SS. Analysis of the reliability of the modified caregiver strain index. J Gerontol B Psychol Sci Soc Sci. 2003 Mar;58(2):S127-32. doi: 10.1093/geronb/58.2.s127. PMID 12646602
- [Result] Fralick M, Bartsch E, Ritchie CS, Sacks CA. Estimating the Use of Potentially Inappropriate Medications Among Older Adults in the United States. J Am Geriatr Soc. 2020 Dec;68(12):2927-2930. doi: 10.1111/jgs.16779. Epub 2020 Aug 25. PMID 32841366
- [Result] Gupta A, Jin G, Reich A, Prigerson HG, Ladin K, Kim D, Ashana DC, Cooper Z, Halpern SD, Weissman JS. Association of Billed Advance Care Planning with End-of-Life Care Intensity for 2017 Medicare Decedents. J Am Geriatr Soc. 2020 Sep;68(9):1947-1953. doi: 10.1111/jgs.16683. Epub 2020 Aug 27. PMID 32853429
- [Result] Alexandre PK, Hwang S, Roth KB, Gallo JJ, Eaton WW. COSTS OF DEPRESSION FROM CLAIMS DATA FOR MEDICARE RECIPIENTS IN A POPULATION-BASED SAMPLE. J Health Hum Serv Adm. 2016 Summer;39(1):72-94. PMID 27483975
- [Result] Subramaniam A, Ueno R, Tiruvoipati R, Darvall J, Srikanth V, Bailey M, Pilcher D, Bellomo R. Defining ICD-10 surrogate variables to estimate the modified frailty index: a Delphi-based approach. BMC Geriatr. 2022 May 13;22(1):422. doi: 10.1186/s12877-022-03063-x. PMID 35562684
- [Result] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Result] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Result] Living Independently with GRACE Commonwealth Fund. Accessed July 20, 2022. https://www.commonwealthfund.org/publications/case-study/2021/oct/living-independently- grace
- [Result] Butler DE, Frank KI, Counsell SR. The GRACE Model. In: Malone ML, Capezuti EA, Palmer RM, eds. Geriatrics Models of Care: Bringing "Best Practice" to an Aging America. Springer International Publishing; 2015:125-138. doi:10.1007/978-3-319-16068-9_10
- [Result] Gruber-Baldini AL, Velozo C, Romero S, Shulman LM. Validation of the PROMIS(R) measures of self-efficacy for managing chronic conditions. Qual Life Res. 2017 Jul;26(7):1915-1924. doi: 10.1007/s11136-017-1527-3. Epub 2017 Feb 26. PMID 28239781
- [Result] PROMIS. Accessed July 20, 2022. https://www.healthmeasures.net/explore-measurement- systems/promis
- [Result] Bickman L, Riemer M, Kelley SD, et al. Peabody Treatment Progress Battery PTPB 2010. Published online 2010:306
- [Result] Scholle SH, Vuong O, Ding L, Fry S, Gallagher P, Brown JA, Hays RD, Cleary PD. Development of and field test results for the CAHPS PCMH Survey. Med Care. 2012 Nov;50 Suppl(Suppl):S2-10. doi: 10.1097/MLR.0b013e3182610aba. PMID 23064272
- [Result] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Result] Shiny CRT Calculator. https://clusterrcts.shinyapps.io/rshinyapp/
- [Result] Accountable Care Organizations (ACOs) CMS. Accessed December 19, 2022. https://www.cms.gov/Medicare/Medicare-Fee-for-Service-Payment/ACO
- [Result] Auerbach DI, Levy DE, Maramaldi P, Dittus RS, Spetz J, Buerhaus PI, Donelan K. Optimal Staffing Models To Care For Frail Older Adults In Primary Care And Geriatrics Practices In The US. Health Aff (Millwood). 2021 Sep;40(9):1368-1376. doi: 10.1377/hlthaff.2021.00401. PMID 34495726
- [Result] McNabney MK, Green AR, Burke M, Le ST, Butler D, Chun AK, Elliott DP, Fulton AT, Hyer K, Setters B, Shega JW. Complexities of care: Common components of models of care in geriatrics. J Am Geriatr Soc. 2022 Jul;70(7):1960-1972. doi: 10.1111/jgs.17811. Epub 2022 Apr 29. PMID 35485287
- [Result] High-Need, High-Cost Patients: Who Are They and How Do They Use Health Care? Commonwealth Fund. Accessed September 3, 2019. https://www.commonwealthfund.org/publications/issue-briefs/2016/aug/high-need-high-cost-patients-who-are-they-and-how-do-they-use
- [Result] Sayer C. "Time Spent at Home" - A Patient-Defined Outcome. NEJM Catalyst. Published online April 26, 2016. Accessed December 21, 2022. https://catalyst.nejm.org/doi/abs/10.1056/CAT.16.0854
- [Result] Shafir A, Garrigues SK, Schenker Y, Leff B, Neil J, Ritchie C. Homebound Patient and Caregiver Perceptions of Quality of Care in Home-Based Primary Care: A Qualitative Study. J Am Geriatr Soc. 2016 Aug;64(8):1622-7. doi: 10.1111/jgs.14244. Epub 2016 Jul 7. PMID 27384919
- [Result] Grant RW, Ashburner JM, Hong CS, Chang Y, Barry MJ, Atlas SJ. Defining patient complexity from the primary care physician's perspective: a cohort study. Ann Intern Med. 2011 Dec 20;155(12):797-804. doi: 10.7326/0003-4819-155-12-201112200-00001. PMID 22184686
- [Result] Weiss KB. Managing complexity in chronic care: an overview of the VA state-of-the-art (SOTA) conference. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):374-8. doi: 10.1007/s11606-007-0379-x. PMID 18026804
- [Result] Feder JL. Predictive modeling and team care for high-need patients at HealthCare Partners. Health Aff (Millwood). 2011 Mar;30(3):416-8. doi: 10.1377/hlthaff.2011.0080. No abstract available. PMID 21383355
- [Result] Conwell LJ, Cohen JW. Characteristics of Persons with High Medical Expenditures in the U.S. Civilian Noninstitutionalized Population, 2002. Published online 2002:6.